Official Study Title: Effects of Boccia Exercises on Upper Extremity Muscle Thickness and Grip

Strength in Hemiparetic Individuals

NCT Number: NCT ID not yet assigned

**Document Type:** Informed voluntary participation form

**Document Date:** 19 November 2025

Principal Investigator: Emre Berk HAZAR

**Institution:** Bayburt University

## INFORMED VOLUNTARY CONSENT FORM

We invite you to participate in the study titled "Examining the Effect of 8-Week Bocce Training on Shoulder and Hand Muscle Architecture in Middle-Aged Individuals Using Ultrasonography and Assessing Some Anthropometric Characteristics." You will be asked to participate in the study for approximately 8 weeks, 3 days a week, for 40 minutes. Participation in this study is entirely voluntary. For the study to achieve its objectives, you are expected to answer all questions completely, sincerely, and provide the answers that best suit you, without being pressured or manipulated by anyone. Reading and approving this form signifies your agreement to participate in the study. However, you have the right not to participate or to withdraw from the study at any time. The information obtained from this study will be used solely for research purposes, and your personal information will be kept confidential. Since personal data will be collected in the study, all necessary measures will be taken to protect personal data in accordance with Law No. 6698 on the Protection of Personal Data and relevant legislation. If you need more information now or later, other than the information provided regarding the purpose of the research, you can ask the researcher now or contact him/her by e-mail at ebhazar@bayburt.edu.tr or by phone at +90 507 031 32 88.

**Subject and Purpose of the Study**: A study will be conducted to examine the effect of 8-week bocce training on shoulder and hand muscle architecture in middle-aged individuals using ultrasonography and to evaluate some anthropometric characteristics.

I have read the information above, which must be provided to participants before the study begins, and I understand the scope and purpose of the study in which I am being asked to participate, as well as my responsibilities as a volunteer. A written and verbal explanation of the study was provided by the researcher identified below. The potential risks and benefits of the study were also explained to me verbally. I was given sufficient assurance that my personal information would be carefully protected.

Under these circumstances, I agree to participate in the research of my own free will, without any pressure or suggestion.

| Participant's: | |
|-----------------------------------------|------------|
| Name-Surname: | |
| Signature: | |
| Contact Information; email: | Telephone: |
| The researcher | |
| Name-Surname: Arş. Gör. Emre Berk HAZAR | |
| Signature: | |